CLINICAL TRIAL: NCT02772666
Title: New Automatic Portable Ophthalmology Device
Brief Title: Novel Portable Diagnostic Device for Automatic Detection of Relative Afferent Pupillary Defect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amirhossein Vejdani, MD, Dr., Mashhad University of Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: IR.MUMS.REC.1395.15
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis; Glaucoma
Keywords: Relative afferent pupillary defect (RAPD); Multiple sclerosis; Glaucoma
MeSH Terms: conditions — Multiple Sclerosis; Glaucoma; Pupil Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- O-Glass (Experimental): All study participants who were diagnosed Relative Afferent Pupillary defect(RAPD) positive according to expert specialist investigations, were enrolled in this study. They were all examined with new device named O-Glass.
  Interventions: Device: O-Glass
- Swinging Flash light Test (Active Comparator): All study participants who were diagnosed Relative Afferent Pupillary defect(RAPD) positive according to expert specialist investigations were also examined with manual diagnostic method, Swinging Flash light Test(SFT). The standard and most common method for Marcus-Gunn test is Swinging Flashlight Test (SFT), which needs a dark room, and the patient will be asked to look toward a distant object, so the pupils are not focused. The patient is asked to gaze into the distance, and the examiner swings the beam of a penlight back and forth from one pupil to the other, and observes the size of pupils and reaction in the eye that is lit.
  Interventions: Other: Swinging Flashlight Test

INTERVENTIONS:
Device: O-Glass — The new diagnostic device to distinguish relative afferent pupillary defect(RAPD).
  Arms: O-Glass
Other: Swinging Flashlight Test — The swinging-flashlight test is used to help a practitioner identify a relative afferent pupillary defect.For an adequate test, vision must not be entirely lost. In dim room light, the examiner notes the size of the pupils. The patient is asked to gaze into the distance, and the examiner swings the beam of a penlight back and forth from one pupil to the other, and observes the size of pupils and reaction in the eye that is lit.
  Other Names: Other diagnostic method
  Arms: Swinging Flash light Test

SUMMARY:
This study is to evaluate the ability of a newly designed device, Optic Nerve Glass (O-Glass) to detect relative afferent pupillary defect (RAPD). In this prospective study, 44 patients (diagnosed RAPD- positive) enrolled the study. They were examined for an RAPD by O-Glass and also manual swinging flashlight method (SFM) . This newly designed instrument captures and records eye pictures. The images will be processed and analyzed using computerized software to calculate pupillary measurements.

DETAILED DESCRIPTION:
Pupil response to light stimulation is a basic clinical approach to the assessment of a patient with visual loss. Asymmetric response may indicate a relative afferent pupillary defect (RAPD). The rapid detection device for relative afferent pupillary defect (present device) is a newly designed portable facility with computerized software on a mobile device. This allows for field ophthalmic examination and identification of RAPDs quickly and accurately and also record pupillary movements for further processing and analysis or send the information and images via Wi-Fi. We aimed at comparing and evaluating this device with available methods to develop a test which is practically easy and quick with objective results and no need for specialist interpretation, so that any technician can perform the test automatically. Distinctive software allows simple use of the device by field personnel with minimal training. Each patient was investigated by swinging flashlight method and the newly constructed automated O-glass. The swinging flashlight test procedure, also called as Marcus Gunn Test, is well known in ophthalmology science.The hardware for this device includes 4 different parts: Camera and optics, light control system, power control system, and the microcontroller.The two main components of the software are the ability to communicate with the hardware wirelessly, and the pattern recognition system.

ELIGIBILITY:
Inclusion Criteria:

* positive relative afferent pupillary defect

Exclusion Criteria:

-

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amirhossein Vejdani, M.D., Study Chair — Mashhad University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided
I have not decided about it.

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: 44 patients diagnosed with relative afferent pupillary defect (RAPD- positive) were enrolled.
Period: O-Glas Then SFT
Arm/Group | All Study Participants
Started | 44
Completed | 44
Not Completed | 0
Period: SFT Then O-Glass
Arm/Group | All Study Participants
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Full Range); unit: years] | 35 [20 to 55]
Gender [Count of Participants; unit: Participants]
  Female | 18
  Male | 26
Region of Enrollment [Number; unit: participants] — Khatam Al-Anbia Eye Hospital, Mashhad, a city in north east of Iran.
  participants
    Iran, Islamic Republic of | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Detected Relative Afferent Pupillary Defect (RAPD)
Description: The instrument illuminated the eyes alternatively and took images and recorded pupillary reflex to this light stimulation.
  All of 44 patients were examined with two methods, SFT and O Glass. SFT method: The well known manual method to diagnose RAPD. O glass method:The device consists of camera and light sources.The red light was on and off for a 5 second interval. Then the white light was on for right eye and 3 seconds later the system captured an image. After 0.5 second the right light was off and the left light turned on, 3 seconds later the image was captured. The images were processed and analyzed using computerized software.
Time Frame: up to 6 months
Measure: Number; unit: participants
Groups:
- O-Glass: 44 patients diagnosed with relative afferent pupillary defect (RAPD- positive) were examined with O-Glass.
- Swinging Flashlight Test: 44 patients diagnosed with relative afferent pupillary defect (RAPD- positive) were examined with manual swinging flashlight test(SFT).
Arm/Group | O-Glass | Swinging Flashlight Test
Number analyzed (Participants) | 44 | 44
participants | 44 | 37

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- All Study Participants: This diagnostic intervention is just an inspection and taking picture of the eye.
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No